CLINICAL TRIAL: NCT02039349
Title: A Novel Compound for Alcoholism Treatment: A Translational Strategy
Brief Title: A Novel Compound for Alcoholism Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of Rhode Island (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 140042; 14-AA-0042
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-12-24

CONDITIONS: Alcoholism; Alcohol-Related Disorders; Alcohol Dependence; Alcohol Drinking Related Problems; Alcohol Drinking
Keywords: Alcoholism; Ghrelin; Ghrelin Antagonism
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Alcohol Drinking | interventions — PF-5190457

INTERVENTIONS:
Drug: PF-05190457

SUMMARY:
Background:

- Hormones are naturally occurring chemicals in your body. Ghrelin is a hormone that is mainly produced by the stomach and stimulates appetite. Some studies suggest it may stimulate alcohol craving and use. Drugs have been developed that block ghrelin. Researchers want to know if people can tolerate a particular drug that blocks ghrelin. It will be given at two dose levels, combined with alcohol.

Objective:

- To determine if a drug that may decrease alcohol consumption when given along with alcohol is safe and tolerable.

Eligibility:

* Healthy adults 21-65 years old who have 14 (women) to 21 (men) drinks a week.
* No one of childbearing potential can participate.

Design:

* Participants will have 3 inpatient clinic visits; each will last 4 days.
* They will have physical exam and blood and urine tests.
* They will have breath tests for alcohol and smoking.
* They will answer health and mood questions.
* Researchers will measure their reaction to smelling alcohol and tasting a sweet drink.
* They will eat only the food provided by the clinic. They will keep a food diary 1 day before each stay.
* They will be randomly assigned to take the study drug or placebo 5 times each stay.
* On Day 3, they will drink alcohol after taking the drug. They will give many blood samples that day through a tube inserted in their skin.
* Smokers can take smoke breaks. Once, they will smoke a cigarette through a device.
* One week after the last stay, participants will have a follow-up visit to answer questions.

DETAILED DESCRIPTION:
Objective: Ghrelin is a 28-aminoacid peptide that stimulates appetite and food intake. It is an endogenous ligand for the growth hormone secretagogue receptor (GHSR1a). Preclinical studies suggest that ghrelin modulates alcohol reward processing. Furthermore, findings from a translational human lab study at Brown University (PI: Leggio) indicate that intravenous (IV) ghrelin administration, compared to placebo, results in an acute increase in craving for alcohol during a cue-reactivity experiment in alcoholic individuals. Therefore, an orally bioavailable, ghrelin receptor antagonist, that can pass through the blood brain barrier holds particular promise as an AD treatment. This project has been recently funded by NCATS. The goals of this protocol are to generate preliminary evidence on the safety and efficacy of a ghrelin receptor antagonist (GHSR1a antagonist), PF-05190457, an existing molecule available under the NIH-Industry Pilot Program at NCATS.

Study population: Non-treatment seeking heavy drinkers (n =20). The study will be conducted in the Inpatient Unit at the NIAAA Intramural Clinical Program.

Study Design: Single-blind dose-escalating placebo-controlled inpatient study using PF-05190457, in non-treatment seeking heavy drinking subjects. This Phase 1b study will be a within-subject design.

Outcome measures: Primary objectives will be to determine: 1) the number of adverse events (AEs) experienced, compared between all three PF-05190457 dose categories (0mg or placebo, 50mg, and 100mg b.i.d.); and 2) the total concentration of the drug, compared between the two non-placebo drug doses (50mg and 100mg b.i.d.), when co-administered with alcohol. We hypothesize that both doses of PF-05190457, as compared to placebo, will not result in an increased number of AEs. As a secondary objective, we will determine whether PF-05190457 dose-dependently affects the subjective effects of alcohol and craving. We will include pharmacokinetics (PK) and pharmacodynamic (PD) investigations conducted at University of Rhode Island (URI; Associate Investigator: Akhlaghi). The PK/PD component will include (i) measuring total, unbound or tissue concentrations of the drug using liquid chromatography tandem mass spectrometry (LC-MS/MS) and evaluation of biomarkers of effect and (ii) estimation of PK and PD parameters by the use of conventional and semi-mechanistic modeling approaches to assist in identifying an optimal dosing regimen of the drug in AD.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males or females 21-65 years old (inclusive);
* Heavy drinking defined as on average at least 21 drinks per week for men or at least 14 drinks for women based on the timeline follow-back (TLFB) done at screening.
* Be in good health as confirmed by medical history, physical examination, ECG, blood/urine lab tests;
* Female subjects must be of non childbearing potential as defined by at least one of the following criteria:

  * Females 45 65 years old, who are menopausal, defined as follows:

    * Females who are between 45 55 years old: they will be considered menopausal if they satisfy all the following three requirements during screening: 1) they are in amenorrhea, defined as absence of menstruation for the previous 12 months; 2) they have a negative urine pregnancy test; and 3) they have a serum FSH level within the laboratory s reference range for postmenopausal females.
    * Females who are between 56 65 years old: they will be considered menopausal if they are in amenorrhea, defined as absence of menstruation for the previous 12 months before screening.
  * OR
  * Females 21-65 years old, who have a documented hysterectomy and/or bilateral oophorectomy.
  * All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy) will be considered to be of childbearing potential.
* Male subjects must use one of the following methods of contraception from the first dose of study medication and until 28 days after dosing:

  * Abstinence.
  * A condom AND one of the following:

    * Vasectomy for more than 6 months.
    * Female partner who meets one of the following conditions:

      * Has had a tubal ligation, hysterectomy, or bilateral oophorectomy;
      * Is post menopausal;
      * Uses one of the following forms of contraception:

        * Copper or hormonal containing IUD;
        * Spermicidal foam/gel/film/cream/suppository;
        * Diaphragm with spermicide;
        * Oral contraceptive;
        * Injectable progesterone;
        * Subdermal implant.

EXCLUSION CRITERIA:

* Interest in receiving treatment for heavy drinking.
* Current DSM-IV diagnosis (based on SCID) of substance dependence (other than alcohol and/or nicotine); a negative urine drug screen will also be required.
* DSM-IV Axis I criteria for a lifetime diagnosis of schizophrenia, bipolar disorder, or other psychoses;
* Active illness within the past 6 months of the screening visit that meet the DSM-IV criteria for a diagnosis of major depressive disorder or anxiety disorder; subjects with a history of attempted suicide will be excluded;
* Clinically significant medical abnormalities (e.g., unstable hypertension, clinically significant EKG abnormalities, Creatinine greater than or equal to 2 mg/dL, liver cirrhosis, AST or ALT > 3x the upper normal limit, hemoglobin <10.5 g/dl);
* Heart rate >100 at screening on two separate measurements given potential of study medication to increase heart rate.
* BMI less than or equal to 18.5 or anorexia given potential of the study medication to reduce appetite.
* BMI greater than or equal to 35 kg/m^2.
* Exclusionary Medications:

  * Naltrexone, acamprosate, alcohol dehydrogenase inhibitors, topiramate, gabapentin, ondansetron, benzodiazepines, beta-blockers, H2-blockers, and alpha-1 blockers, baclofen, and barbiturates as well as hormone replacement therapy; medications and dietary/herbal supplements (like St. John's wort) that interact with Cytochrome P450 3A4. All of the medications in the previous sentence will not be allowed if they have been taken within 2 weeks of study medication administration.
  * PF-05190457 is a substrate for P-glycoproteins (P-gp or encoded by ABCB1 gene) based on information from in vitro or animal models. Patients that are required to take the following inhibitors and inducers of P-gp are excluded unless the subject stops taking these agents for 2 weeks for P-gp inhibitors or 6 weeks for P-gp inducers before study medication administration.

Inhibitors: Amiodarone, azithromycin, captopril, carvedilol, clarithromycin, conivaptan, cyclosporine, diltiazem, dronedarone, erythromycin, felodipine, itraconazole, ketoconazole, lopinavir and ritonavir, quercetin, quinidine, ranolazine, verapamil

Inducers: Avasimibe, carbamazepine, phenytoin, rifampin, St John s wort, tipranavir/ritonavir [From Drug Development and Drug Interactions: Table of Substrates, Inhibitors and Inducers, table 12, from http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm#substrates]

* History of epilepsy or alcohol-related seizures;
* patients who have diabetes and/or are treated with any drug with glucose lowering properties such as sulfonylurea, insulin, metformin, thiazolidinediones (TZD), Dipeptidyl peptidase-4(DPP4) inhibitors, or Glucagon-like peptide-1(GLP-1)agonists (due to the glucose-lowering properties of PF-05190457 observed in healthy volunteers);
* History of alcohol-induced flushing reactions.
* Clinically significant alcohol withdrawal symptoms, as assessed by a CIWA-Ar score > 8 at screening.
* Any other reason or clinical condition for which the PI or the MAI will consider unsafe for a possible participant to participate in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01-03; Primary Completion 2015-10-01 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Side effects/adverse events and maximum tolerated dose of PF-05190457 alone and in combination with alcohol administration. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Leggio L, Schwandt ML, Oot EN, Dias AA, Ramchandani VA. Fasting-induced increase in plasma ghrelin is blunted by intravenous alcohol administration: a within-subject placebo-controlled study. Psychoneuroendocrinology. 2013 Dec;38(12):3085-91. doi: 10.1016/j.psyneuen.2013.09.005. Epub 2013 Sep 13. PMID 24090583
- [Background] Leggio L, Ferrulli A, Cardone S, Nesci A, Miceli A, Malandrino N, Capristo E, Canestrelli B, Monteleone P, Kenna GA, Swift RM, Addolorato G. Ghrelin system in alcohol-dependent subjects: role of plasma ghrelin levels in alcohol drinking and craving. Addict Biol. 2012 Mar;17(2):452-64. doi: 10.1111/j.1369-1600.2010.00308.x. Epub 2011 Mar 11. PMID 21392177
- [Background] Leggio L, Zywiak WH, Fricchione SR, Edwards SM, de la Monte SM, Swift RM, Kenna GA. Intravenous ghrelin administration increases alcohol craving in alcohol-dependent heavy drinkers: a preliminary investigation. Biol Psychiatry. 2014 Nov 1;76(9):734-41. doi: 10.1016/j.biopsych.2014.03.019. Epub 2014 Mar 25. PMID 24775991
- [Background] Leggio L. Role of the ghrelin system in alcoholism: Acting on the growth hormone secretagogue receptor to treat alcohol-related diseases. Drug News Perspect. 2010 Apr;23(3):157-66. doi: 10.1358/dnp.2010.23.3.1429490. PMID 20440417
- [Background] Bhattacharya SK, Andrews K, Beveridge R, Cameron KO, Chen C, Dunn M, Fernando D, Gao H, Hepworth D, Jackson VM, Khot V, Kong J, Kosa RE, Lapham K, Loria PM, Londregan AT, McClure KF, Orr ST, Patel J, Rose C, Saenz J, Stock IA, Storer G, VanVolkenburg M, Vrieze D, Wang G, Xiao J, Zhang Y. Discovery of PF-5190457, a Potent, Selective, and Orally Bioavailable Ghrelin Receptor Inverse Agonist Clinical Candidate. ACS Med Chem Lett. 2014 Feb 24;5(5):474-9. doi: 10.1021/ml400473x. eCollection 2014 May 8. PMID 24900864
- [Derived] Cobbina E, Lee MR, Leggio L, Akhlaghi F. A Population Pharmacokinetic Analysis of PF-5190457, a Novel Ghrelin Receptor Inverse Agonist in Healthy Volunteers and in Heavy Alcohol Drinkers. Clin Pharmacokinet. 2021 Apr;60(4):471-484. doi: 10.1007/s40262-020-00942-7. Epub 2020 Nov 5. PMID 33155163
- [Derived] Lee MR, Farokhnia M, Cobbina E, Saravanakumar A, Li X, Battista JT, Farinelli LA, Akhlaghi F, Leggio L. Endocrine effects of the novel ghrelin receptor inverse agonist PF-5190457: Results from a placebo-controlled human laboratory alcohol co-administration study in heavy drinkers. Neuropharmacology. 2020 Jun 15;170:107788. doi: 10.1016/j.neuropharm.2019.107788. Epub 2019 Sep 23. PMID 31557492
- [Derived] Denney WS, Sonnenberg GE, Carvajal-Gonzalez S, Tuthill T, Jackson VM. Pharmacokinetics and pharmacodynamics of PF-05190457: The first oral ghrelin receptor inverse agonist to be profiled in healthy subjects. Br J Clin Pharmacol. 2017 Feb;83(2):326-338. doi: 10.1111/bcp.13127. Epub 2016 Oct 29. PMID 27621150